CLINICAL TRIAL: NCT02583412
Title: Preparedness for and Response to Meningococcal Outbreaks: a Pilot Study of the Immunogenicity, Reactogenicity and Tolerability of Two Schedules of a 4CmenB Vaccine in Adolescents and Young Adults
Brief Title: Pilot Study of the Immunogenicity, Reactogenicity and Tolerability of Two Schedules of a 4CmenB Vaccine in Adolescents and Young Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: University of British Columbia (Other); University of Calgary (Other); Université de Montréal (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Joanne Langley, Principal Investigator, Canadian Immunization Research Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CT11
Record Dates: First submitted 2015-09-04; First posted 2015-10-22 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Meningococcal Serogroup B
MeSH Terms: interventions — 4CMenB vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: Accelerated Schedule (Active Comparator)
  Interventions: Biological: Bexsero®; Biological: Havrix®
- Group 2: Standard Schedule (Active Comparator)
  Interventions: Biological: Bexsero®; Biological: Havrix®

INTERVENTIONS:
Biological: Bexsero® — Multicomponent meningococcal B vaccine
Biological: Havrix® — Hepatitis A vaccine

SUMMARY:
The overall aim of this study is to determine if an accelerated "Bexsero® (Multicomponent meningococcal B vaccine)" schedule compared to a standard schedule is immunogenic, safe, and tolerable, in order to increase capacity for rapid outbreak control. In this pilot study no formal hypothesis is tested.

DETAILED DESCRIPTION:
A pilot study to evaluate the feasibility of a rapid clinical trial at the time of a meningococcal B outbreak, comparing an accelerated schedule of 4CMen B (0, 3 weeks) to the 0, 2 months schedule, to determine if the more compressed schedule is immunogenic, safe and tolerable. A shorter schedule offers the potential benefit of more rapid direct and indirect protection, and use of fewer public health resources for implementation.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 17 to 25 years.
* Current or intended student at an educational setting in the 2015-2016 year.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Significant renal or hepatic impairment.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participant in another research trial involving an investigational product or medical device in the prior 12 weeks.
* Previous bacteriologically confirmed N. meningitidis disease.
* Prior receipt of a meningococcal B vaccine
* Hypersensitivity to any vaccine component of products used in this study (see product monographs)
* Immunodeficiency or autoimmune disease

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Immune responses to 4CMenB vaccine, as measured by human Serum Bactericidal Assay (hSBA | Baseline to day 180
  Immune responses will be measured:
  * Prior to 4CMenB vaccine (baseline)
  * To a single dose of 4CMenB vaccine 21 days post-immunization
  * 21 days after the second dose of an accelerated compared to a standard 4CMenB schedule
  * Six months after an accelerated 4CMenB vaccine schedule and a standard schedule

SECONDARY OUTCOMES:
Number of solicited general adverse events | Day 0-6
  The number of participants in each vaccine group with each symptom day 0 to 6 after vaccine will be summarized. Each vaccine participant will record if they had any symptoms (yes/no) and the severity (mild, moderate, or severe.)
  The following general AEs will be solicited:
  * Drowsiness
  * Fever
  * Nausea
  * Diarrhea
  * Vomiting
  * Generalized muscle aches
Number of unsolicited general adverse events | Day 0-21
  The number of participants in each vaccine group with each symptom day 0 to 21 after vaccine will be summarized. Each vaccine participant will record if they had any symptoms (yes/no) and the severity (mild, moderate, or severe.)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 reported in the accelerated vaccine schedule compared to a standard schedule | From injection to Day 180
Number of solicited local and systemic injections site reactions | Day 0-6
  The following local (injection-site) AEs will be solicited:
  * Pain at injection site
  * Redness at injection site
  * Swelling at injection site

CONTACTS AND LOCATIONS:
Overall Officials: Joanne M Langley, MD, MSc, FRCPC, Principal Investigator — IWK Health Centre, Dalhousie University
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Sharkey K, Beernink PT, Langley JM, Gantt S, Quach C, Dold C, Liu Q, Galvan M, Granoff DM. Anti-Factor H Antibody Reactivity in Young Adults Vaccinated with a Meningococcal Serogroup B Vaccine Containing Factor H Binding Protein. mSphere. 2019 Jul 3;4(4):e00393-19. doi: 10.1128/mSphere.00393-19. PMID 31270173